CLINICAL TRIAL: NCT07166809
Title: The Effect of Dynamic Neuromuscular Stabilization-Based Training Combined With Pelvic Floor Muscle Training on Lower Urinary Tract Symptoms and Pelvic Floor Functions in Women With Multiple Sclerosis
Brief Title: The Effect of DNS-Based Training Combined With PFMT on LUTS and Pelvic Floor Functions in Women With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Seda Kilic, Lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/554
Record Dates: First submitted 2025-08-27; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Women With Multiple Sclerosis; Multiple Sclerosis; Lower Urinary Track Symptoms; Pelvic Floor Disorder
Keywords: Multiple sclerosis; Lower urinary tract symptoms; Pelvic floor muscle training; stabilization; Dynamic neuromuscular stabilization
MeSH Terms: conditions — Multiple Sclerosis; Pelvic Floor Disorders; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: pelvic floor muscle training (PFMT) only or PFMT combined with Dynamic Neuromuscular Stabilization (DNS). Both groups followed an 8-week program, with the intervention group receiving additional supervised DNS exercises.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFMT (Active Comparator): Participants in the PFMT group received only an 8-week remotely monitored pelvic floor muscle training program without additional DNS-based exercises.
  Interventions: Other: Pelvic Floor Muscle Training (PFMT)
- PFMT+DNS (Experimental): Participants in the PFMT+DNS group received the same 8-week remotely monitored pelvic floor muscle training program, in addition to supervised Dynamic Neuromuscular Stabilization exercises three times per week.
  Interventions: Other: Pelvic Floor Muscle Training (PFMT); Other: Pelvic Floor Muscle Training combined with Dynamic Neuromuscular Stabilization (PFMT+DNS)

INTERVENTIONS:
Other: Pelvic Floor Muscle Training (PFMT) — A structured pelvic floor muscle training program delivered remotely for 8 weeks, including exercises designed to strengthen and improve the endurance, coordination, and control of the pelvic floor muscles.
  Other Names: PFMT
Other: Pelvic Floor Muscle Training combined with Dynamic Neuromuscular Stabilization (PFMT+DNS) — Participants received the same 8-week remotely monitored pelvic floor muscle training program as the PFMT group, in addition to supervised Dynamic Neuromuscular Stabilization exercises three times per week. DNS exercises aimed to enhance core stability, postural control, and coordination to support pelvic floor muscle function.
  Other Names: PFMT+DNS
  Arms: PFMT+DNS

SUMMARY:
The goal of this randomized controlled trial is to investigate whether adding Dynamic Neuromuscular Stabilization (DNS)-based training to Pelvic Floor Muscle Training (PFMT) can improve lower urinary tract symptoms (LUTS) and pelvic floor functions in women with multiple sclerosis (MS), aged 28-54 years.

The main questions it aims to answer are:

Does DNS combined with PFMT improve lower urinary tract symptoms more effectively than PFMT alone?

Does DNS combined with PFMT enhance pelvic floor muscle function more effectively than PFMT alone?

Researchers will compare PFMT alone versus PFMT combined with DNS-based stabilization exercises to see if DNS provides additional benefits.

Participants will:

Perform an 8-week remotely monitored Pelvic Floor Muscle Training program.

In the DNS+PFMT group, complete supervised Dynamic Neuromuscular Stabilization exercises three times a week.

Undergo assessments including:

Urinary Symptom Profile questionnaire and uroflowmetry for objective evaluation of lower urinary tract symptoms,

International Consultation on Incontinence Questionnaire-Short Form,

Overactive Bladder Questionnaire (8-item version),

Vaginal palpation using the PERFECT (Power, Endurance, Repetitions, Fast contractions, Every Contraction Timed) scheme,

Electromyography (muscle electrical activity measurement) for pelvic floor muscles,

Magnetic Resonance Imaging (MRI) for diaphragm function evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Diagnosis of multiple sclerosis with an Expanded Disability Status Scale (EDSS) score below 6
* Pelvic floor muscle strength greater than grade 1 according to the Modified Oxford Scale (MOS)
* No pelvic floor muscle training received in the previous six months

Exclusion Criteria:

* Multiple sclerosis relapse within the past month
* Pregnant or within six months postpartum
* Diagnosis of urinary tract infection
* Any medical condition that could interfere with participation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants who self-identify as women are eligible to participate.
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Lower urinary tract symptoms (LUTS) severity | Baseline and 8 weeks after intervention
  Lower urinary tract symptoms (LUTS) severity measured by the Urinary Symptom Profile (USP) questionnaire. The USP includes three subdomains: stress urinary incontinence (0-9), overactive bladder symptoms (0-21), and voiding symptoms (0-9) with total scores ranging from 0 to 39, higher scores indicating greater severity.
Urinary incontinence severity and impact on quality of life | baseline and 8 weeks
  Urinary incontinence severity and impact on quality of life assessed by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). The ICIQ-SF assesses urinary leakage frequency, volume, and daily life impact, scored 0-21, with ≥8 indicating clinically significant incontinence (Cronbach's α = 0.71).
Overactive bladder symptoms | Baseline and 8 weeks
  Overactive bladder symptoms measured by the Overactive Bladder-Version 8 (OAB-V8). The OAB-V8 comprises eight 5-point items (total 0-40), with higher scores reflecting greater bother, and a cutoff of 11 indicating clinically relevant overactive bladder symptoms
Objective urinary flow parameters | Baseline and 8 weeks
  Objective urinary flow parameters assessed by uroflowmetry. Uroflowmetry, a non-invasive diagnostic test, was performed. Participants were instructed to void naturally into a uroflowmeter device in a private setting. The device automatically recorded maximum bladder capacity (mL), maximum flow rate (Qmax, mL/s), average flow rate (Qavg, mL/s), and voided volume (mL).
Pelvic Floor Muscle Function - Vaginal Palpation | Baseline and 8 weeks
  Pelvic floor muscle function was assessed by digital vaginal palpation using the PERFECT scheme. The examiner inserted one or two gloved fingers into the vagina and instructed the participant to contract and relax the pelvic floor muscles. Parameters recorded included: Power (maximum voluntary contraction, graded on the Modified Oxford Scale), Endurance (duration of sustained contraction in seconds), Repetitions (number of sustained contractions), Fast contractions (number of quick contractions), and Every Contraction Timed (consistency of contraction timing).
Pelvic floor muscle function - Electromyography (EMG) | Baseline and 8 weeks
  EMG biofeedback device was used to measure the bioelectrical activity of the pelvic floor muscles. EMG provides an objective evaluation of muscle contraction and relaxation. Intravaginal probes were used as they are considered the gold standard (17). Assessments were performed using the Neurotrac MyoPlus Pro (Verity Medical Ltd.), which recorded parameters such as muscle strength, endurance, relaxation ability, and resting tone. During the EMG evaluation, participants were positioned supine in lithotomy, and a personalized intravaginal probe was inserted by the clinician. After ensuring the participant understood how to correctly contract the pelvic floor muscles, the EMG protocol included a warm-up phase with five contractions and five relaxations, followed by three cycles of 5-second contraction and 5-second relaxation periods.

SECONDARY OUTCOMES:
Diaphragm Function - Magnetic Resonance Imaging (MRI) | Baseline and 8 weeks
  Diaphragm function was assessed using Magnetic Resonance Imaging (MRI). Dynamic MRI sequences were performed during inspiration and expiration to evaluate diaphragm mobility and muscle activity. Measurements included excursion (movement in millimeters) and changes in diaphragm thickness as indicators of contractile function.
Perceived level of improvement - Global Perceived Effect Scale (GPE) | Baseline and 8 weeks
  The Global Perceived Effect Scale (GPE) was used to assess participants' perceived level of improvement following the intervention. This validated questionnaire categorizes perceived recovery into nine levels, ranging from (1) "very much improved" to (9) "very much worse," with intermediate options such as "moderately improved" or "unchanged."
Treatment adherence - Visual Analog Scale (VAS) | Baseline and 8 weeks
  Treatment adherence was evaluated using a Visual Analog Scale (VAS). Participants rated their adherence to the treatment program on a scale from 0 to 10, where 0 indicated "not adherent at all" and 10 indicated "completely adherent."

CONTACTS AND LOCATIONS:
Overall Officials: SEDA KILIC, DR., Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis Üniversitesi, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including questionnaire scores (Urinary Symptom Profile, International Consultation on Incontinence Questionnaire-Short Form, Overactive Bladder Questionnaire), pelvic floor muscle function assessments (PERFECT scheme and electromyography), demographic information (age), and group assignment, will be shared. All data will be anonymized to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Available 12 months after publication of the main study results
Access Criteria: De-identified individual participant data and supporting documents (Study Protocol, Statistical Analysis Plan, Informed Consent Form, Analytic Code) will be available to qualified researchers for academic and scientific purposes. Researchers must submit a request to the Principal Investigator with a brief research proposal. Access will be granted after approval and signing a data use agreement. Data will be shared through a secure repository to ensure confidentiality.